# **CLINICAL STUDY PROTOCOL**

A Placebo-Controlled, Double-Blind, Randomized, Phase 2 Study to Evaluate the Effect of Obicetrapib 10 mg Daily in Combination With Ezetimibe 10 mg Daily as an Adjunct to High-Intensity Statin Therapy: The ROSE 2 Study

**Investigational Product:** Obicetrapib **Protocol Number:** TA-8995-202

## **Sponsor:**

NewAmsterdam Pharma BV
Gooimeer 2-35
1411 DC
Naarden
The Netherlands

Telephone: +31 35 699 30 00 Fax: +31 20 240 07 79

Version Number: 1.0 Date: 16 September 2021

## **Confidentiality Statement**

The information in this document is confidential and is not to be disclosed without the written consent of NewAmsterdam Pharma BV except to the extent that disclosure would be required by law and for the purpose of evaluating and/or conducting a clinical study for NewAmsterdam Pharma BV. You are allowed to disclose the contents of this document only to your Institutional Review Board and study personnel directly involved with conducting this protocol. Persons to whom the information is disclosed must be informed that the information is confidential and proprietary to NewAmsterdam Pharma BV and that it may not be further disclosed to third parties.

NCT number: NCT05266586

This NCT number has been applied to the document for the purposes of posting on clinicaltrials.gov

# **SIGNATURE PAGE**

STUDY TITLE: A Placebo-Controlled, Double-Blind, Randomized, Phase 2 Study to Evaluate the Effect of Obicetrapib 10 mg Daily in Combination With Ezetimibe 10 mg Daily as an Adjunct to High-Intensity Statin Therapy: The ROSE 2 Study



## INVESTIGATOR AGREEMENT

By signing below I agree that:

I have read this protocol. I approve this document and I agree that it contains all necessary details for carrying out the study as described. I will conduct this study in accordance with the design and specific provision of this protocol and will make a reasonable effort to complete the study within the time designated. I will provide copies of this protocol and access to all information furnished by NewAmsterdam Pharma BV to study personnel under my supervision. I will discuss this material with them to ensure they are fully informed about the study drug and study procedures. I will let them know that this information is confidential and proprietary to NewAmsterdam Pharma BV and that it may not be further disclosed to third parties. I understand that the study may be terminated or enrollment suspended at any time by NewAmsterdam Pharma BV, with or without cause, or by me if it becomes necessary to protect the best interests of the study participants.

I agree to conduct this study in full accordance with Food and Drug Administration Regulations, Institutional Review Board Regulations, and International Council for Harmonisation Guidelines for Good Clinical Practices.

| Investigator's Signature | <br>Date |
|-----------------------------|----------|
| Investigator's Printed Name | |

## **SYNOPSIS**

**TITLE:** A Placebo-Controlled, Double-Blind, Randomized, Phase 2 Study to Evaluate the Effect of Obicetrapib 10 mg Daily in Combination With Ezetimibe 10 mg Daily as an Adjunct to High-Intensity Statin Therapy: The ROSE 2 Study

PROTOCOL NUMBER: TA-8995-202

**INVESTIGATIONAL PRODUCT:** Obicetrapib

PHASE: 2

**INDICATION:** Dyslipidemia

#### **OBJECTIVES:**

The primary objective of this study is to evaluate the effect of objectrapib 10 mg + ezetimibe 10 mg combination therapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on low-density lipoprotein cholesterol (LDL-C) at Day 84.

The secondary objectives of this study include the following, in hierarchical order:

- To evaluate the effect of obicetrapib 10 mg monotherapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on LDL-C at Day 84;
- To evaluate the effect of obicetrapib 10 mg + ezetimibe 10 mg combination therapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on apolipoprotein B (ApoB) at Day 84; and
- To evaluate the effect of obicetrapib 10 mg monotherapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on ApoB at Day 84.

The exploratory objectives of this study include the following:

- To evaluate the effect of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy, when used as an adjunct to high-intensity statin therapy, on non-high-density lipoprotein cholesterol (non-HDL-C), very low-density lipoprotein cholesterol (VLDL-C), high-density lipoprotein (HDL) cholesterol (HDL-C), triglycerides (TG), apolipoprotein E (ApoE), lipoprotein (a) (Lp[a]), and HDL-ApoE at Day 84;
- To evaluate the effect of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy, when used as an adjunct to high-intensity statin therapy, on the proportion of participants achieving predefined LDL-C targets at Day 84;

- To assess the mean trough plasma levels of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy at steady state on Days 28, 84, and 112; and
- To evaluate the safety and tolerability profiles of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy, when used as an adjunct to high-intensity statin therapy, assessed by clinical laboratory values and incidence of adverse events (AEs).

#### **POPULATION:**

The population for this study includes men and women 18 to 75 years of age, inclusive, with a body mass index <40 kg/m², fasting LDL-C levels >70 mg/dL, and TG levels <400 mg/dL at the Screening Visit, who are currently receiving high-intensity statin therapy.

#### STUDY DESIGN AND DURATION:

This study will be a placebo-controlled, double-blind, randomized, Phase 2 study to evaluate the efficacy, safety, and tolerability of obicetrapib 10 mg, both in combination with ezetimibe 10 mg and as monotherapy, as an adjunct to high-intensity statin therapy. This study will take place at approximately 20 sites in the United States.

# Screening Period

At the Screening Visit, participants will be required to sign an informed consent form (ICF) before any study-related procedures are performed. After signing the ICF, participants will be assessed for study eligibility.

## **Treatment Period**

Up to 2 weeks after the Screening Visit, participants will return to the site on Day 1 (Visit 2) and confirm study eligibility before being randomized and beginning treatment. Approximately 114 eligible participants (38 participants per treatment group) will be randomized in a 1:1:1 ratio to 1 of the following treatment groups:

- Combination therapy: Obicetrapib 10 mg + ezetimibe 10 mg (administered as one 10 mg obicetrapib tablet and one 10 mg ezetimibe capsule);
- Obicetrapib monotherapy: Obicetrapib 10 mg (administered as one 10 mg obicetrapib tablet and 1 placebo capsule); or
- Placebo (administered as 1 placebo tablet and 1 placebo capsule).

During the 12-week Treatment Period, the assigned study drugs will be administered by the participants orally with water, once daily on Day 1 to Day 84 at approximately the same time each morning. Participants will return to the site on Day 28 (±2 days), Day 84 (±2 days), and Day 112 (±2 days) for efficacy, safety, and pharmacokinetic (PK) assessments. Participants, Investigators, the Clinical Research Organization, and the Sponsor will be blinded to all lipid results from Day 1 (Visit 2) for the first participant until all enrolled participants complete the Day 84 (End of Treatment) visit or are withdrawn from the study, in order to protect blinding to treatment assignment.

## Safety Follow-Up Period

Participants will return to the site for a Safety Follow-up Visit (Visit 5) approximately 4 weeks after the end of the Treatment Period for safety and PK assessments.

## DOSAGE FORMS AND ROUTE OF ADMINISTRATION:

The study drugs include obicetrapib 10 mg, ezetimibe 10 mg, and matching placebo for each. Participants will be randomized to receive combination therapy (obicetrapib 10 mg + ezetimibe 10 mg [administered as one 10 mg obicetrapib tablet and one 10 mg ezetimibe capsule]); obicetrapib monotherapy (obicetrapib 10 mg [administered as one 10 mg obicetrapib tablet and 1 placebo capsule]), or placebo (administered as 1 placebo tablet and 1 placebo capsule) on Day 1 to Day 84. Study drugs (1 tablet and 1 capsule) will be administered by the participant orally with water, once daily on Day 1 to Day 84 at approximately the same time each morning.

#### **EFFICACY VARIABLES:**

The primary efficacy endpoint is the percent change from Day 1 to Day 84 in LDL-C for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group.

The secondary efficacy endpoints include the following, in hierarchical order:

- Percent change from Day 1 to Day 84 in LDL-C for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group;
- Percent change from Day 1 to Day 84 in ApoB for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group; and
- Percent change from Day 1 to Day 84 in ApoB for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group.

The exploratory efficacy endpoints include the following:

- Percent change from Day 1 to Day 84 in non-HDL-C, VLDL-C, HDL-C, TG, ApoE, Lp(a), and HDL-ApoE for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group and for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group; and
- Proportion of participants at Day 84 that achieve LDL-C <2.6 mmol/L (<100 mg/dL), LDL-C <1.8 mmol/L (<70 mg/dL), and LDL-C <1.3 mmol/L (<50 mg/dL) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group and for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group.</li>

## PHARMACOKINETIC VARIABLES:

Plasma obicetrapib concentrations, both in combination with ezetimibe and as monotherapy, will be assessed at the scheduled PK collection times.

## **SAFETY VARIABLES:**

The safety and tolerability profile of obicetrapib 10 mg, both in combination with ezetimibe 10 mg and as monotherapy, will be assessed by clinical laboratory assessments (chemistry and hematology), vital signs, physical examinations, and the incidence of AEs.

## **STATISTICAL ANALYSES:**

A Statistical Analysis Plan (SAP) will be finalized before database lock. Any changes to the methods described in the SAP will be described and justified as needed in the Clinical Study Report. All study-collected data will be summarized by treatment group using descriptive statistics, graphs, and/or raw data listings. Descriptive statistics for continuous variables will include number of participants (n), mean, standard deviation (SD), median, minimum, and maximum values. Analysis of categorical variables will include frequency and percentage.

# **Analysis Populations**

The Intent-to-Treat (ITT) Population will include all participants randomized into the study. Treatment classification will be based on the randomized treatment.

The Modified ITT (mITT) Population will include all participants in the ITT Population who receive at least 1 dose of any study drug and have a baseline value for the LDL-C assessment. Any efficacy measurement obtained during the Safety Follow-up Visit (Visit 5) after a participant permanently discontinues the study drug or after a participant receives an excluded medication and/or procedure will be removed from the mITT analysis. Treatment classification will be based on the randomized treatment. The mITT Population will be used for the primary analysis of all efficacy endpoints.

The Per-Protocol (PP) Population will include all participants in the mITT Population who have a baseline value for the LDL-C assessment, have a Day 84 value for the LDL-C assessment, and who do not experience a major protocol deviation that could potentially impact the primary efficacy endpoint. The PP Population, along with the reason for exclusion, will be finalized prior to study unblinding.

The PK Population will include all participants in the mITT Population who have sufficient blood samples collected for valid estimation of PK parameters.

The Safety Population will include all participants who receive at least 1 dose of any study drug. Treatment classification will be based on the actual treatment received. The Safety Population will be the primary population used for the safety analyses.

# Analysis of Efficacy

The mITT Population will be the primary population for the efficacy analyses. Efficacy will also be analyzed using the ITT Population and the PP Population as supportive analyses.

The primary efficacy analysis of the percent change from Day 1 to Day 84 in LDL-C will be performed using a mixed model for repeated measures (MMRM) approach. The analysis will include fixed effects for treatment, visit, and treatment-by-visit interaction, along with a covariate of the baseline value as a continuous covariate. The Restricted Maximum Likelihood estimation approach will be used with an unstructured covariance matrix. The least squares means, standard errors, and 2-sided 95% confidence intervals for the combination group and for comparison of the

combination treatment group to the placebo group will be provided. Sensitivity analyses for various assumptions of missing data will be imputed using multiple imputation methodology. Results will be combined using Rubin's method. Full details of the model(s) and imputation will be provided in the SAP.

Similar MMRM models will be developed to examine the secondary efficacy endpoints. In order to maintain the overall Type I error rate, the secondary efficacy endpoints will be tested sequentially at the 0.05 significance level according to the order of hierarchy specified above.

Similar MMRM models will be used for the percent change from Day 1 to Day 84 in non-HDL-C, VLDL-C, HDL-C, TG, ApoE, Lp(a), and HDL-ApoE.

The proportion of participants at Day 84 that achieve LDL-C <2.6 mmol/L (<100 mg/dL), LDL-C <1.8 mmol/L (<70 mg/dL), and LDL-C <1.3 mmol/L (<50 mg/dL) will be examined through logistic regression models for binary variables with covariants of the treatment groups and the baseline variable.

No adjustment will be made for multiplicity in testing the exploratory efficacy endpoints. Nominal p-values will be provided when applicable. Any additional sensitivity and/or supplemental analyses will be defined in the SAP.

## Analysis of Pharmacokinetics

Plasma obicetrapib concentrations will be summarized with descriptive statistics based on the PK Population. Exploration of any relationships with obicetrapib exposure will be performed, as appropriate.

# **Analysis of Safety**

The Safety Population will be the primary population for the safety analyses. All safety endpoints will be summarized descriptively. No statistical inference will be applied to the safety endpoints.

## **SAMPLE SIZE DETERMINATION:**

A sample size of at least 108 evaluable participants (ie, 36 participants per treatment group) will provide >90% power to detect a 30% difference in LDL-C reduction at Day 84 (SD of 15%) for each of the obicetrapib treatment groups compared with the placebo group at a 1-sided significance level of 0.025.

The sample size for this study was determined in order to provide sufficient power for the analyses of the primary and first secondary efficacy endpoints described above. Therefore, assuming an approximately 5% dropout rate, enrollment of approximately 114 participants (ie, 38 participants per treatment group) is planned for this study. This sample size will also contribute sufficient participant exposure and safety data.

Participants will be stratified according to their Screening Visit LDL-C levels (≥100 or <100 mg/dL).

**SITES:** Approximately 20 sites in the United States

# **SPONSOR:**

NewAmsterdam Pharma BV Gooimeer 2-35 1411 DC Naarden The Netherlands

Telephone: +31 35 699 30 00

Fax: +31 20 240 07 79

# TABLE OF CONTENTS

| Si | gnatur | e Page | | 2 |
|---|---|---|---|---|
| In | vestiga | ator Ag | reement | 3 |
| Sy | nopsis | S | | 4 |
| Та | ble of | Conter | nts | 10 |
| Li | st of A | bbrevia | ations and Definition of Terms | 14 |
| 1 | Introduction and Background Information | | | 16 |
| | 1.1 | Chole | steryl Ester Transfer Protein Inhibitors | 16 |
| | 1.2 | Obice | trapib (TA-8995) | 17 |
| | 1.3 | 1.3 Clinical Development of Obicetrapib | | 17 |
| | 1.4 | Rationale | | 18 |
| | | 1.4.1 | Rationale for Obicetrapib and Ezetimibe Combination Therapy | 18 |
| | | 1.4.2 | Dose Selection Rationale for Obicetrapib | 19 |
| | 1.5 | Risk/I | Benefit | 19 |
| | | 1.5.1 | Coronavirus Disease 2019 Impacts | 19 |
| 2 | Study Objectives | | | 21 |
| | 2.1 | 1 Primary Objective | | |
| | 2.2 | 2.2 Secondary Objectives | | 21 |
| | 2.3 | 8 Exploratory Objectives | | |
| 3 | Study Description | | | 22 |
| | 3.1 | Summ | nary of Study Design | 22 |
| | | 3.1.1 | Screening Period | 22 |
| | | 3.1.2 | Treatment Period | 22 |
| | | 3.1.3 | Safety Follow-Up Period. | 22 |
| | | 3.1.4 | Coronavirus Disease 2019 Contingency Measures | 22 |
| | 3.2 | Study | Indication | 23 |
| 4 | Selection and Withdrawal of Participants | | | 24 |
| | 4.1 | 4.1 Inclusion Criteria | | 24 |
| | 4.2 | .2 Exclusion Criteria | | |
| | 4.3 | Retesting | | |
| | 4.4 | 4 Rescreening | | |

| | 4.5 | Withd | lrawal Criteria | 26 |
|---|---|---|---|---|
| 5 | Stud | tudy Treatments | | |
| | 5.1 | 1 Treatment Groups | | |
| | 5.2 | Rationale for Dosing | | 27 |
| | 5.3 | Randomization and Blinding | | 27 |
| | 5.4 | .4 Breaking the Blind | | |
| | 5.5 | 5 Drug Supplies | | 28 |
| | | 5.5.1 | Formulation and Packaging | 28 |
| | | 5.5.2 | Study Drug Preparation and Dispensing | 29 |
| | | 5.5.3 | Study Drug Administration | 29 |
| | | 5.5.4 | Treatment Compliance | 29 |
| | | 5.5.5 | Storage and Accountability | 30 |
| | 5.6 | Prior a | and Concomitant Medications and/or Procedures | 30 |
| | | 5.6.1 | Excluded Medications and/or Procedures | 30 |
| | | 5.6.2 | Allowed Medications and/or Procedures | 30 |
| | | 5.6.3 | Documentation of Prior and Concomitant Medication Use | 30 |
| 6 | Stud | y Proce | dures | 31 |
| 7 | Efficacy and Pharmacokinetic Assessments | | | 32 |
| | 7.1 | 1 Efficacy Assessments | | |
| | 7.2 | Pharm | nacokinetic Assessments | 32 |
| | 7.3 | Serum | Archive Sample | 33 |
| 8 | Safety Assessments 3- | | | 34 |
| | 8.1 | Adver | se Events | 34 |
| | | 8.1.1 | Adverse (Drug) Reaction | 35 |
| | | 8.1.2 | Unexpected Adverse Drug Reaction | 35 |
| | | 8.1.3 | Assessment of Adverse Events by the Investigator | 35 |
| | 8.2 | Seriou | as Adverse Events | 36 |
| | 8.3 | Serious Adverse Event Reporting – Procedures for Investigators | | 37 |
| | 8.4 | Pregnancy Reporting | | |
| | 8.5 | Expedited Reporting | | |
| | 8.6 | Special Situation Reports | | 38 |
| | 8.7 | Clinic | al Laboratory Evaluations | 39 |

| | | 8.7.1 | Chemistry and Hematology Assessments | 39 |
|---|---|---|---|---|
| | | 8.7.2 | Endocrinology Assessments | 39 |
| | | 8.7.3 | Aldosterone Assessment | 39 |
| | 8.8 | 8.8 Vital Signs | | 39 |
| | 8.9 | Weight and Height | | 40 |
| | 8.10 | Demog | graphics | 40 |
| | 8.11 | 8.11 Electrocardiograms | | 40 |
| | 8.12 Physical Examinations | | al Examinations | 40 |
| 9 | Statis | stics | | 41 |
| | 9.1 | Analys | sis Populations | 41 |
| | 9.2 | Statist | ical Methods | 41 |
| | | 9.2.1 | Analysis of Efficacy | 41 |
| | | | 9.2.1.1 Primary efficacy analysis | 41 |
| | | | 9.2.1.2 Secondary efficacy analyses | 42 |
| | | | 9.2.1.3 Exploratory analyses | 42 |
| | | 9.2.2 | Analysis of Pharmacokinetics | 42 |
| | | 9.2.3 | Analysis of Safety | 42 |
| | | 9.2.4 | Interim Analysis | 42 |
| | | 9.2.5 | Sample Size Determination | 42 |
| 10 Data Management and Record Keeping | | | 44 | |
| | 10.1 | Data N | Management | 44 |
| | | 10.1.1 | Data Handling | 44 |
| | | 10.1.2 | Computer Systems. | 44 |
| | | 10.1.3 | Data Entry | 44 |
| | | 10.1.4 | Medical Information Coding. | 44 |
| | | 10.1.5 | Data Validation | 44 |
| | 10.2 | Record | l Keeping | 44 |
| | 10.3 | End of | Study | 45 |
| 11 | Inves | tigator | Requirements and Quality Control | 46 |
| | 11.1 | Ethica | Conduct of the Study | 46 |
| | 11.2 | Institu | tional Review Board | 46 |
| | 11.3 | Inform | ed Consent | 46 |

# NewAmsterdam Pharma BV Clinical Study Protocol TA-8995-202

| 11.4 Study Monitoring Requirements | 46 |
|------------------------------------------|----|
| 11.5 Disclosure of Data | 47 |
| 11.6 Retention of Records | 47 |
| 11.7 Publication Policy | 47 |
| 11.8 Financial Disclosure | 48 |
| 12 Study Administrative Information | 49 |
| 12.1 Protocol Amendments | 49 |
| 13 References | 50 |
| Appendix A: Schedule of Procedures | 51 |
| Appendix B: Clinical Laboratory Analytes | 53 |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | Adverse event |
| ApoA1 | Apolipoprotein A1 |
| ApoB | Apolipoprotein B |
| ApoE | Apolipoprotein E |
| ASCVD | Atherosclerotic cardiovascular disease |
| CETP | Cholesteryl ester transfer protein |
| COVID-19 | Coronavirus Disease 2019 |
| CRA | Clinical Research Associate |
| CRO | Clinical Research Organization |
| CV | Cardiovascular |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EDC | Electronic data capture |
| EIU | Exposure In Utero |
| FDA | Food and Drug Administration |
| FSH | Follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| HbA1c | Glycosylated hemoglobin |
| HDL | High-density lipoprotein |
| HDL-C | High-density lipoprotein cholesterol |
| HMGCR | 3-hydroxy-3-methylglutaryl-coenzyme A reductase |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation |
| IRB | Institutional Review Board |
| IRT | Interactive response technology |
| ITT | Intent-to-Treat |
| LDL | Low-density lipoprotein |
| LDL-C | Low-density lipoprotein cholesterol |
| Lp(a) | Lipoprotein (a) |
| mITT | Modified Intent-to-Treat |
| MMRM | Mixed model for repeated measures |
| non-HDL-C | Non-high-density lipoprotein cholesterol |
| PCSK9 | Proprotein convertase subtilisin kexin type 9 |
| PK | Pharmacokinetic(s) |
| PP | Per-Protocol |
| QTc | Heart rate-corrected QT interval |
| QTcF | Heart rate-corrected QT interval using Fridericia's formula |

| Abbreviation | Definition |
|--------------|-----------------------------------------------|
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TG | Triglyceride(s) |
| ULN | Upper limit of normal |
| VLDL-C | Very low-density lipoprotein cholesterol |
| WHO | World Health Organization |

#### 1 INTRODUCTION AND BACKGROUND INFORMATION

Dyslipidemias are disorders of lipoprotein metabolism, including lipoprotein overproduction or deficiency, which may be manifested by elevation of the levels of the serum total cholesterol, low-density lipoprotein (LDL) cholesterol (LDL-C) and triglyceride (TG) concentrations, and a decrease in the levels of high-density lipoprotein (HDL) cholesterol (HDL-C) concentration. These disorders are generally diagnosed by measuring the serum lipids and classified by the pattern of elevation/reduction in the lipid/lipoprotein fractions. Dyslipidemia itself does not generally cause any symptoms, but it can lead to symptomatic vascular disease including coronary artery disease and peripheral arterial disease. It is acknowledged that while there are a number of genetic and lifestyle factors which contribute to the development of vascular disease, dyslipidemia is 1 of the most prominent risk factors and normalization of the lipid profile has been a major target in cardiovascular (CV) protection strategies.<sup>1</sup>

Statins are generally the drug of first choice in treating dyslipidemia. Statins are considered as the most potent, most effective, and best tolerated drugs for reducing LDL-C levels. Many patients, despite treatment with high-intensity statin therapy, do not achieve acceptable levels of LDL-C with statins alone.

There is a need for chronic therapies which will robustly reduce elevated LDL-C levels when used adjunctive to high-intensity statin therapy.

# 1.1 Cholesteryl Ester Transfer Protein Inhibitors

Cholesteryl ester transfer protein (CETP) is a plasma glycoprotein produced in the liver and adipose tissue. It circulates in the blood, bound primarily to HDL-C, and is involved in the transfer of cholesteryl esters and TG between lipoproteins. In particular, it mediates the transfer of cholesteryl esters from HDL to apolipoprotein B (ApoB)-containing particles, eg, very low-density lipoprotein and LDL-C, in exchange for TG. As a result, cholesteryl ester from HDL can be taken up by the liver through scavenger receptor class B type 1; this action also leads to decreased HDL-C and ultimately to increased LDL-C.

Inhibition of CETP activity reduces ApoB and LDL-C and increases HDL-C. CETP-inhibiting therapies were originally developed based on the premise that increasing HDL-C levels would prevent CV events. However, clinical study results and Mendelian randomization data have revealed that these effects are caused by changes in the concentration of ApoB-containing particles (including LDL particles) rather than changes in the HDL-C levels.<sup>2,3</sup> Therefore, the LDL-C and ApoB-lowering effects, which arise from CETP inhibition and occur through upregulation of the LDL receptor, will benefit patients with elevated LDL-C and increased CV risk.

Ference and colleagues have recently investigated the association between changes in LDL-C levels (and other lipoproteins) and the risk of CV events related to variants in the CETP gene alone and in combination with variants in the 3-hydroxy-3-methylglutaryl-coenzyme A reductase (HMGCR) gene.<sup>2</sup> The results of these Mendelian randomization analyses demonstrate that treatment with a CETP inhibitor has the potential to effectively reduce the risk of CV events. Both genetic and therapeutic inhibition of CETP leads to quantitatively concordant changes in LDL-C and ApoB levels. A further Mendelian randomization analysis concluded that the clinical benefit of lower LDL-C levels per unit difference may specifically be related to the absolute reduction in ApoB-containing lipoprotein particles.<sup>4</sup>

# 1.2 Obicetrapib (TA-8995)

Obicetrapib (TA-8995) is a selective CETP inhibitor. Inhibition of CETP by obicetrapib blocks the transfer of cholesteryl ester from non-atherogenic HDL particles to particles in lipoprotein fractions (including LDL) that cause atherosclerosis and reduces the concentration of cholesterol in LDL, as well as other atherogenic lipoproteins. Obicetrapib also has several additional compound-specific activities that are hypothesized to be beneficial in patients. In a recent study, obicetrapib treatment not only reduced the number of ApoB-containing particles that constitute LDL-C, it also increased apolipoprotein E (ApoE), which led to the removal of cholesterol via the liver and also reduced lipoprotein (a) (Lp[a]).<sup>5</sup> Finally, obicetrapib not only potently increases HDL-C and the concentration of apolipoprotein A1 (ApoA1)-containing lipoproteins but has been demonstrated to be a potent inducer of cholesterol efflux, which is the main driver of reverse cholesterol transport.<sup>6</sup> This effect is considered important because it is expected to reduce established atheroma burden.

# 1.3 Clinical Development of Obicetrapib

Both single ascending dose (TA-8995-01) and multiple ascending dose (TA-8995-02) studies of obicetrapib have been conducted in healthy volunteers. A formal, thorough QT/QTc study (TA-8995-04) demonstrated that obicetrapib has no effect on the QTcF. A drug-drug interaction study (TA-8995-05) showed no significant effect of obicetrapib on P-glycoprotein activity, but showed that obicetrapib is a mild inducer of cytochrome P450 3A4. A mass balance study in healthy males concluded that obicetrapib is steadily absorbed, and the principal route of excretion was in the feces (TA-8995-07). Finally, bioequivalence between obicetrapib capsule and tablet formulations was investigated (TA-8995-08).

The first patient study conducted was a Phase 2 clinical study (TA-8995-03) in Denmark and The Netherlands where the aim was to evaluate the optimal dose of obicetrapib alone and in combination with statins in patients with mild dyslipidemia. This study concluded that a 10 mg daily dose of obicetrapib therapy resulted in an LDL-C reduction of 45.4%, an HDL-C increase of 179.0%, an ApoA1 increase of 63.4%, and a significant increase of HDL-C efflux capacity. Furthermore, given on top of atorvastatin 20 mg, obicetrapib 10 mg resulted in an additional 50.3% reduction in LDL-C. A second patient study (TA-8995-06) showed a statistically significant reduction in Lp(a) levels following 12 weeks of obicetrapib treatment.

Two Phase 2 studies of obicetrapib (TA-8995-303 and TA-8995-201) are currently nearing completion. The first study, TA-8995-303, is evaluating the LDL-lowering effects of obicetrapib 5 mg in combination with ezetimibe 10 mg in participants with mild dyslipidemia. The second study, TA-8995-201, is evaluating the LDL-lowering effects of obicetrapib (both 5 mg and 10 mg) as an adjunct to high intensity statin therapy in participants with dyslipidemia who are on high-intensity statins.

Two Phase 3 studies of obicetrapib 10 mg investigating the treatment of elevated LDL-C levels in participants with established atherosclerotic CV disease (ASCVD), as well as heterozygous familial hypercholesterolemia, are currently in development. One study (TA-8995-301) will include participants on maximally tolerated lipid-lowering therapy, including maximally tolerated doses of statins with an LDL-C inclusion criterion of ≥100 mg/dL. The other study (TA-8995-302) will also include participants who are on maximally tolerated lipid-lowering therapy, including maximally tolerated doses of statins with an LDL-C inclusion criterion of ≥70 mg/dL and

<100 mg/dL. Together, these 2 pivotal studies will evaluate the effects of obicetrapib 10 mg in populations requiring further LDL-C reduction across a range of baseline LDL-C values relevant to contemporary clinical practice.

A third Phase 3 study (TA-8995-304) will investigate the effect of obicetrapib 10 mg on clinical outcomes (ie, major adverse CV events, including CV death, non-fatal myocardial infarction, non-fatal stroke, or non-elective coronary revascularization).

#### 1.4 Rationale

Chronic LDL-C elevation leads to progressive accumulation of arterial atherosclerotic lesions that require long-term management. While lifestyle changes are the primary intervention, these measures seldom reduce plasma LDL-C by more than 15%, and pharmacologic treatments are required to adequately treat hyperlipidemia.<sup>7</sup>

Statins are considered as first-line therapy for reducing LDL-C levels. However, despite lipid lowering therapy with statins, many patients are unable to achieve acceptable levels of LDL-C.

Proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitors are one alternative to statins. However, there are several limitations with these therapies, including high costs, limited long-term outcome data relative to statins, and muscle-related events. In addition, because PCSK9 inhibitors are injectable, this poses a less attractive option for patients who prefer oral medications.

Accordingly, there remains an unmet need for therapies to effectively reduce elevated LDL-C levels and CV risk at an acceptable cost, a convenient dosage form, and a more favorable safety profile to encourage long-term use and patient compliance. Obicetrapib, an oral CETP inhibitor, has demonstrated safety and efficacy in the reduction of LDL-C, in addition to other beneficial effects. The combination of obicetrapib and ezetimibe, an oral cholesterol absorption inhibitor, could be a valuable alternative to a PCSK9 inhibitor in patients who require additional LDL-C lowering despite high-intensity statin therapy.

## 1.4.1 Rationale for Obicetrapib and Ezetimibe Combination Therapy

Ezetimibe selectively inhibits intestinal cholesterol absorption. Ezetimibe used as monotherapy for patients with hypercholesterolemia significantly reduces serum LDL-C levels, as evidenced by a meta-analysis of 8 randomized, double-blind, placebo-controlled studies, with a statistically significant mean reduction in LDL-C of 18.58% compared with placebo.<sup>8</sup> Ezetimibe in combination with statin therapy further reduces LDL-C levels. A meta-analysis of 27 studies, including more than 21,000 patients, demonstrated a 15.1% greater reduction in LDL-C in patients treated with statin and ezetimibe in combination compared with statin alone.<sup>9</sup> The IMPROVE-IT study,<sup>10</sup> in which simvastatin 40 mg daily was compared with a combination of simvastatin 40 mg plus ezetimibe 10 mg in 18,144 patients with acute coronary syndrome, demonstrated a modest but statistically significant further reduction in future CV events (a 2% absolute risk reduction over 7 years) in the combination group compared with statins alone. These large long-term studies have also demonstrated an excellent safety profile for ezetimibe. Importantly, additional Mendelian randomization studies have revealed that the CETP inhibitor HMGCR inhibitor interaction does not occur when a CETP inhibitor is combined with ezetimibe.

A Phase 2 study is currently underway evaluating the LDL-lowering effects of obicetrapib 5 mg in combination with ezetimibe 10 mg in participants with mild dyslipidemia and no prior CV events (TA-8995-303).

To evaluate the potential of a higher dose of obicetrapib in combination with ezetimibe to augment reduction in LDL-C and ApoB, this study will evaluate the effect of obicetrapib 10 mg in combination with ezetimibe 10 mg in participants currently receiving high-intensity statin therapy (atorvastatin 40 or 80 mg or rosuvastatin 20 or 40 mg) as part of their guideline-directed medical therapy.

# 1.4.2 Dose Selection Rationale for Obicetrapib

In clinical studies in healthy volunteers, obicetrapib was generally well tolerated in single doses up to 150 mg and multiple doses up to 25 mg/day for 21 days. In clinical studies in patients, obicetrapib was also well tolerated after daily dosing of 10 mg for 12 weeks, both alone and in combination with 2 different statins. Near maximal effects were observed with the 10 mg obicetrapib dose. At this dose level, CETP activity and concentrations were reduced, HDL-C levels were increased, and LDL-C levels were decreased. There were no dose-related adverse events (AEs) identified and no clinically significant changes in vital signs, electrocardiograms (ECGs), or hematology or biochemistry parameters in any clinical studies. A statistically significant reduction in Lp(a) levels from baseline was also observed at the 10 mg obicetrapib dose level. Therefore, the present study will utilize a dose of 10 mg obicetrapib in participants with ASCVD who are not adequately controlled despite maximally tolerated lipid-modifying therapies.

#### 1.5 Risk/Benefit

The primary pharmacology in in vitro, ex vivo, and in vivo studies have demonstrated that obicetrapib has the ability to inhibit CETP, decrease LDL-C levels, increase HDL-C levels, and importantly, reduce the number of atherogenic ApoB-containing particles in a way that is useful in the treatment of dyslipidemia.

The safety pharmacology studies have demonstrated that obicetrapib has no adverse effect on critical physiological systems (eg, central nervous system, respiratory system, gastric emptying, urinary tract, and steroidal hormonal production [including aldosterone levels]) at doses up to 300 mg/kg in rats.

In clinical studies in patients, obicetrapib was also well tolerated after daily dosing of 10 mg for 12 weeks, both alone and in combination with 2 different statins. There were no dose-related AEs identified and no clinically significant changes in vital signs, ECGs, or hematology or biochemistry parameters in any clinical studies.

## 1.5.1 Coronavirus Disease 2019 Impacts

In March 2020, the Coronavirus Disease 2019 (COVID-19), caused by infection with severe acute respiratory syndrome coronavirus 2, was characterized as a pandemic by the World Health Organization (WHO). The COVID-19 pandemic has impacted clinical studies worldwide due to quarantines, site closures, travel limitations, diversion of resources, and/or general interruptions in study-related procedures. This study will be initiated during the ongoing COVID-19 pandemic. The Sponsor has reviewed guidance from regulatory authorities and reports from the literature while planning study start-up and conduct (ie, Food and Drug Administration [FDA] 2020).<sup>11</sup>

The Sponsor will communicate with sites before study initiation and during the conduct of the study concerning the potential impact of COVID-19 on study-related procedures and overall conduct. The Sponsor will continue to monitor COVID-19 activity in the geographic areas and

institutions where the trial will be conducted and conduct an ongoing risk assessment throughout the study. The risk assessment will be documented on an ongoing basis in the Sponsor's trial master file.

This study protocol includes contingency measures to ensure participant safety while enabling sites to generate reliable data and maintain integrity of the study and study data (see Section 3.1.4). The impacts of these implemented contingency measures on the outcomes of this study, including any protocol deviations that result from COVID-19 illness and/or COVID-19 control measures, will be discussed in the Clinical Study Report.

Treatment with standard of care and/or emergency use authorization medications, including vaccinations and boosters, for COVID-19 will be permitted during this study. There is no known negative impact of vaccination on obicetrapib efficacy and safety, nor any known negative impact of obicetrapib on vaccination efficacy and safety.

#### 2 STUDY OBJECTIVES

# 2.1 Primary Objective

The primary objective of this study is to evaluate the effect of objectrapib 10 mg + ezetimibe 10 mg combination therapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on LDL-C at Day 84.

# 2.2 Secondary Objectives

The secondary objectives of this study include the following, in hierarchical order:

- To evaluate the effect of obicetrapib 10 mg monotherapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on LDL-C at Day 84;
- To evaluate the effect of obicetrapib 10 mg + ezetimibe 10 mg combination therapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on ApoB at Day 84; and
- To evaluate the effect of obicetrapib 10 mg monotherapy compared with placebo, when used as an adjunct to high-intensity statin therapy, on ApoB at Day 84.

# 2.3 Exploratory Objectives

The exploratory objectives of this study include the following:

- To evaluate the effect of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy, when used as an adjunct to high-intensity statin therapy, on non-high-density lipoprotein cholesterol (non-HDL-C), very low-density lipoprotein cholesterol (VLDL-C), HDL-C, TG, ApoE, Lp(a), and HDL-ApoE at Day 84;
- To evaluate the effect of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy, when used as an adjunct to high-intensity statin therapy, on the proportion of participants achieving predefined LDL-C targets at Day 84;
- To assess the mean trough plasma levels of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy at steady state on Days 28, 84, and 112; and
- To evaluate the safety and tolerability profiles of obicetrapib 10 mg + ezetimibe 10 mg combination therapy and obicetrapib 10 mg monotherapy, when used as an adjunct to high-intensity statin therapy, assessed by clinical laboratory values and incidence of AEs.

## 3 STUDY DESCRIPTION

# 3.1 Summary of Study Design

This study will be a placebo-controlled, double-blind, randomized, Phase 2 study to evaluate the efficacy, safety, and tolerability of obicetrapib 10 mg, both in combination with ezetimibe 10 mg and as monotherapy, as an adjunct to high-intensity statin therapy. This study will take place at approximately 20 sites in the United States.

## 3.1.1 Screening Period

At the Screening Visit, participants will be required to sign an informed consent form (ICF) before any study-related procedures are performed. After signing the ICF, participants will be assessed for study eligibility.

## 3.1.2 Treatment Period

Up to 2 weeks after the Screening Visit, participants will return to the site on Day 1 (Visit 2) and confirm study eligibility before being randomized and beginning treatment. Approximately 114 eligible participants (38 participants per treatment group) will be randomized in a 1:1:1 ratio to 1 of the following treatment groups:

- Combination therapy: Obicetrapib 10 mg + ezetimibe 10 mg (administered as one 10 mg obicetrapib tablet and one 10 mg ezetimibe capsule);
- Obicetrapib monotherapy: Obicetrapib 10 mg (administered as one 10 mg obicetrapib tablet and 1 placebo capsule); or
- Placebo (administered as 1 placebo tablet and 1 placebo capsule).

During the 12-week Treatment Period, the assigned study drugs will be administered by the participants orally with water, once daily on Day 1 to Day 84 at approximately the same time each morning. Participants will return to the site on Day 28 (±2 days), Day 84 (±2 days), and Day 112 (±2 days) for efficacy, safety, and pharmacokinetic (PK) assessments. Participants, Investigators, the Clinical Research Organization (CRO), and the Sponsor will be blinded to all lipid results from Day 1 (Visit 2) for the first participant until all enrolled participants complete the Day 84 (End of Treatment) visit or are withdrawn from the study, in order to protect blinding to treatment assignment.

## 3.1.3 Safety Follow-Up Period

Participants will return to the site for a Safety Follow-up Visit (Visit 5) approximately 4 weeks after the end of the Treatment Period for safety and PK assessments.

## 3.1.4 Coronavirus Disease 2019 Contingency Measures

In cases of COVID-19 limitations, it is the Investigator's responsibility to assure the safety of participants. If necessary, the Sponsor will implement and document mitigation strategies. At the Investigator's discretion, the study visit(s) can be conducted in-clinic or virtually. If conducted virtually, the visit will include alternative methods for safety, efficacy, and distribution/collection of study drug, including but not limited to phone/video contact, alternative location for biologic

sample collection, alternative secure delivery of study drug, home health care (if available), and a secured way of transferring participant data from and to home health services and the site.

If these contingency measures occur, the Sponsor will document the changes made, communicate recommendations about such changes in a timely fashion to minimize or prevent disruptions to the study, and support sites in implementing these changes. Documentation of these cases and the site's management of participants should be recorded in the Investigator study files. In the absence of a COVID-19 impact, it is expected that Investigators and participants follow the protocol requirements as set forth.

# 3.2 Study Indication

The indication for this study is dyslipidemia.

#### 4 SELECTION AND WITHDRAWAL OF PARTICIPANTS

## 4.1 Inclusion Criteria

Participants who meet all of the following criteria will be eligible to participate in the study:

- 1. Understanding of the study procedures, willingness to adhere to the study schedules, and agreement to participate in the study by giving written informed consent prior to screening procedures;
- 2. Men or women 18 to 75 years of age, inclusive, at the Screening Visit;
  - Women may be enrolled if all 3 of the following criteria are met:
    - They are not pregnant;
    - They are not breastfeeding; and
    - They do not plan on becoming pregnant during the study.
  - Women of childbearing potential must have a negative urine pregnancy test at the Screening Visit. Note: Women are not considered to be of childbearing potential if they meet 1 of the following criteria as documented by the Investigator:
    - They have had a hysterectomy or tubal ligation at a minimum of 1 cycle prior to signing the ICF; or
    - They are postmenopausal, defined as ≥1 year since their last menstrual period for women ≥55 years of age or ≥1 year since their last menstrual period and have a follicle-stimulating hormone (FSH) level in the postmenopausal range for women <55 years of age.</p>
  - O Women of childbearing potential must agree to use an effective method of avoiding pregnancy from screening to 90 days after the last visit. Men whose partners are of childbearing potential must agree to use an effective method of avoiding pregnancy from screening to 90 days after the last visit. Effective methods of avoiding pregnancy are contraceptive methods with a Pearl index of <1 used consistently and correctly (including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, diaphragm with spermicide, male or female condoms with spermicide, or cervical cap) or a sterile sexual partner.
- 3. Fasting LDL-C levels >70 mg/dL and TG levels <400 mg/dL at the Screening Visit; and
- 4. Currently receiving high-intensity statin therapy (atorvastatin 40 or 80 mg or rosuvastatin 20 or 40 mg) at a stable dose for 8 weeks prior to screening and intending to remain at the same stable dose throughout the study duration.

## 4.2 Exclusion Criteria

Participants who meet any of the following criteria will be excluded from participation in the study:

- 1. Body mass index  $\ge 40 \text{ kg/m}^2$  at the Screening Visit;
- 2. Current clinically significant CV disease, including but not limited to:
  - Major adverse CV event within 3 months prior to randomization; or
     Note: A major adverse CV event is defined as CV death, non-fatal myocardial infarction, non-fatal stroke, or non-elective coronary revascularization.
  - o New York Heart Association Functional Classification Class III or IV heart failure.
- 3. Glycosylated hemoglobin (HbA1c) ≥10% at the Screening Visit;
- 4. Uncontrolled hypertension, ie, sitting systolic blood pressure >160 mmHg and/or sitting diastolic blood pressure >90 mmHg. One retest will be allowed, at which point if the retest result is no longer exclusionary, the participant may be randomized;
- 5. Active muscle disease or persistent creatine kinase concentration >3 × the upper limit of normal (ULN). One retest will be allowed after 1 week to verify the result, at which point if the retest result is no longer exclusionary, the participant may be randomized;
- 6. Estimated glomerular filtration rate <60 mL/min, calculated using the Chronic Kidney Disease Epidemiology Collaboration equation; 12
- 7. Hepatic dysfunction as evidenced by any laboratory abnormality as follows: gamma-glutamyl transferase, alanine aminotransferase, or aspartate aminotransferase >2 × ULN, or total bilirubin >1.5 × ULN:
- 8. Anemia, defined as hemoglobin concentration <11 g/dL for men and hemoglobin concentration <9 g/dL for women;
- 9. History of malignancy within 5 years prior to screening, with the exception of non-melanoma skin cancers;
- 10. History of alcohol and/or drug abuse within 5 years prior to screening;
- 11. Treatment with other investigational products or devices within 30 days or 5 half-lives, whichever is longer, prior to screening;
- 12. History of participation in any clinical trial evaluating obicetrapib;
- 13. Treatment with any PCSK9 inhibitor within 10 weeks prior to randomization or bempedoic acid within 2 weeks prior to randomization;
- 14. Evidence of any other clinically significant, non-cardiac disease or condition that, in the opinion of the Investigator, would preclude participant in the study; or
- 15. Known CETP inhibitor allergy or intolerance.

## 4.3 Retesting

If laboratory abnormalities during screening are considered by the Investigator to be transient, then the laboratory tests may be repeated once during screening. The Investigator's rationale for retesting should be documented. If the retest result is no longer exclusionary, the participant may be randomized.

# 4.4 Rescreening

A participant who is screened and does not meet the study eligibility criteria may be considered for rescreening upon Sponsor and/or Medical Monitor consultation and approval. Rescreened participants will be assigned a new participant number. Rescreening should occur no less than 5 days after the last Screening Visit.

#### 4.5 Withdrawal Criteria

Participation in this study may be discontinued for any of the following reasons:

- The participant withdraws consent or requests discontinuation from the study for any reason;
- Occurrence of any medical condition or circumstance that exposes the participant to substantial risk and/or does not allow the participant to adhere to the requirements of the protocol;
- Any serious AE (SAE), clinically significant AE, severe laboratory abnormality, intercurrent illness, or other medical condition, which indicates to the Investigator that continued participation is not in the best interest of the participant;
- Pregnancy;
- Requirement of prohibited concomitant medication;
- Participant failure to comply with protocol requirements or study-related procedures; or
- Termination of the study by the Sponsor or the regulatory authority.

Unless the participant withdraws consent, participants who discontinue study drug early should be encouraged to complete the full panel of assessments scheduled for the Early Termination Visit promptly and complete a Safety Follow-up Visit (Visit 5) 4 weeks after the last dose of study drug. PK samples will not be collected during the Safety Follow-up Visit for participants who discontinue study drug early without withdrawing consent or for participants who withdraw prematurely from the study. The reason for participant withdrawal must be documented in the electronic case report form (eCRF).

In the case of a participant lost to follow-up, attempts to contact the participant must be made and documented in the participant's medical records.

Withdrawn participants will not be replaced.

#### 5 STUDY TREATMENTS

# 5.1 Treatment Groups

Participants will be randomized in a 1:1:1 ratio to 1 of the following treatment groups:

- Combination therapy: Obicetrapib 10 mg + ezetimibe 10 mg (administered as one 10 mg obicetrapib tablet and one 10 mg ezetimibe capsule);
- Obicetrapib monotherapy: Obicetrapib 10 mg (administered as one 10 mg obicetrapib tablet and 1 placebo capsule); or
- Placebo (administered as 1 placebo tablet and 1 placebo capsule).

# 5.2 Rationale for Dosing

In clinical studies in healthy volunteers, obicetrapib was generally well tolerated in single doses up to 150 mg and multiple doses up to 25 mg/day for 21 days. In clinical studies in patients, obicetrapib was also well tolerated after daily dosing of 10 mg for 12 weeks, both alone and in combination with 2 different statins. Near maximal effects were observed with the 10 mg obicetrapib dose. At this dose level, CETP activity and concentrations were reduced, HDL-C levels were increased, and LDL-C levels were decreased. There were no dose-related AEs identified and no clinically significant changes in vital signs, ECGs, or hematology or biochemistry parameters in any clinical studies. A statistically significant reduction in Lp(a) levels from baseline was also observed at the 10 mg obicetrapib dose level. Therefore, the present study will utilize a dose of 10 mg obicetrapib in participants with ASCVD who are not adequately controlled despite maximally tolerated lipid-modifying therapies.

The ezetimibe dose of 10 mg is the current FDA-approved dose.

# 5.3 Randomization and Blinding

Participants who meet all eligibility criteria will be randomized into the study. Participants will be randomized in a 1:1:1 ratio to receive combination therapy (obicetrapib 10 mg + ezetimibe 10 mg [administered as one 10 mg obicetrapib tablet and one 10 mg ezetimibe capsule]), obicetrapib monotherapy (obicetrapib 10 mg [administered as one 10 mg obicetrapib tablet and 1 placebo capsule]); or placebo (administered as 1 placebo tablet and 1 placebo capsule).

At randomization, participants will be stratified according to their Screening Visit LDL-C level (≥100 or <100 mg/dL). An automated interactive response technology (IRT) system will be used to assign the participant to 1 of the 3 treatment groups.

Participants, Investigators, the CRO, and the Sponsor will be blinded to all lipid results from Day 1 (Visit 2) for the first participant until all enrolled participants complete the Day 84 (End of Treatment) visit or are withdrawn from the study, in order to protect blinding to treatment assignment.

# 5.4 Breaking the Blind

Unblinding by request of an Investigator should occur only in the event of an emergency or AE, for which it is necessary to know the study drugs to determine an appropriate course of therapy for the participant. If the Investigator or qualified designee must identify the treatment assignment of

an individual participant, the Investigator or qualified designee should request the treatment assignment from the IRT system. The Investigator is advised not to reveal the treatment assignment to other sites or Sponsor personnel.

Prior to unblinding, and if the situation allows, the Investigator should consult with the Sponsor's Medical Monitor. If this is impractical, the Investigator must notify the Sponsor's Medical Monitor as soon as possible, without revealing the treatment assignment of the unblinded participant. The Investigator must document the participant identification and the date and time for breaking the blind and must clearly explain the reasons for breaking the blind.

Medically necessary care should not be delayed for unblinding information (ie, the Investigator should treat the participant based on the participant's signs/symptoms without waiting for the unblinding process to be completed).

For participants who are unblinded and withdrawn from the study, study staff should make every effort to complete the full panel of assessments scheduled for the Early Termination Visit and complete a Safety Follow-up Visit (Visit 5) 4 weeks after the last dose.

## 5.5 Drug Supplies

## 5.5.1 Formulation and Packaging

The study drugs consist of 10 mg obicetrapib tablets or matching placebo tablets and over-encapsulated 10 mg ezetimibe tablets or matching placebo capsules. All study drugs are manufactured in accordance with International Council for Harmonisation (ICH) current Good Manufacturing Practice.

Obicetrapib tablets are round, white film-coated tablets, with no identifying markings, containing 10 mg of obicetrapib calcium drug substance.

Placebo tablets for obicetrapib are matching round, white film-coated tablets, with no identifying markings.

Ezetimibe capsules are 10 mg ezetimibe tablets filled into capsule shells, 1 tablet per capsule. Each capsule also contains an excipient material, common to the tablets, as a filler to prevent the tablet from rattling in the capsule shell.

Placebo capsules to match the ezetimibe capsules are the identical capsule shells filled with the excipient filler material only (no tablets).

Obicetrapib and placebo tablets and ezetimibe and placebo capsules will be packaged into kits providing the 2 study drugs for each treatment group. The kits will be clearly labelled to indicate which tablets/capsules to use on each day. Each kit will provide a sufficient supply for 28 days of dosing, with enough for an extra 4 days of dosing in case the participant needs to postpone the next visit. The shelf-life will be assigned based on the stability of the individual study drugs and will not be greater than the expiry date of the input ezetimibe tablets. The kits will be stored below 25°C.

The physical, chemical, and pharmaceutical formulation properties and characteristics of the obicetrapib tablets are described in the Investigator's Brochure.

All study drugs will be labelled in accordance with all applicable local regulatory requirements.

# 5.5.2 Study Drug Preparation and Dispensing

The study drugs include obicetrapib 10 mg, ezetimibe 10 mg, and matching placebo for each. Participants will be randomized to receive combination therapy (obicetrapib 10 mg + ezetimibe 10 mg [administered as one 10 mg obicetrapib tablet and one 10 mg ezetimibe capsule]); obicetrapib monotherapy (obicetrapib 10 mg [administered as one 10 mg obicetrapib tablet and 1 placebo capsule]), or placebo (administered as 1 placebo tablet and 1 placebo capsule) on Day 1 to Day 84. Study drugs (1 tablet and 1 capsule) will be administered by the participant orally with water, once daily on Day 1 to Day 84 at approximately the same time each morning.

At Visit 2 (Day 1), participants will receive 1 kit (containing 32 obicetrapib tablets or matching placebo tablets and 32 ezetimibe capsules or matching placebo capsules totaling 64 tablets/capsules per kit) with the study drugs appropriate for the participant's treatment group. At Visit 3 (Day 28), participants will receive 2 kits as described above. Each kit will provide a sufficient supply for 28 days of dosing, with enough for an extra 4 days of dosing in case the participant needs to postpone the next visit. Participants will be instructed to take 2 units from the kit each day. The kit will be clearly labelled to indicate which tablets/capsules to use on each day. Participants will be instructed to bring all unused study drugs to the site at the next visit.

This study protocol includes contingency measures to manage disruptions due to COVID-19 control measures, including modifications to study drug dispensation specific to situations where COVID-19 is impacting study conduct. See Section 3.1.4 for details of COVID-19 contingency measures. In the absence of a COVID-19 impact, it is expected that Investigators and participants follow the protocol requirements as set forth.

## 5.5.3 Study Drug Administration

Study drugs (1 tablet and 1 capsule) will be administered by the participant orally with water, once daily on Day 1 to Day 84 at approximately the same time each morning. On days with visits scheduled, study drugs should be administered with water following all fasted blood samples. At Visits 3 and 4, participants will dose from the kit received at the previous visit (Visits 2 and 3, respectively).

If a participant forgets to take study drug on a given day, they should take the next dose as normal and should not take a double dose to make up for the forgotten dose.

## 5.5.4 Treatment Compliance

Compliance to the study drug regimen will be evaluated by counting unused tablets and capsules. Participants will be instructed to bring all unused study drugs to the site at Visits 3 and 4. During the Treatment Period, if compliance is not between 80% and 120%, inclusive, the participant will be counselled about the importance of compliance to the regimen. If the limits are exceeded at 2 consecutive visits, a decision will be made by the Investigator and Sponsor as to whether the participant should be withdrawn from the study.

# 5.5.5 Storage and Accountability

All study drugs must be stored below 25°C (77°F) in a secure area with access limited to the Investigator and authorized site personnel.

In accordance with regulatory requirements, the Investigator or designated site personnel must document the amount of study drug dispensed and/or administered to participants, the amount returned by participants, and the amount received from and returned to the Sponsor (or representative) when applicable. Study drug accountability records must be maintained throughout the course of the study. The accountability unit for this study is a tablet or capsule. Discrepancies are to be reconciled or resolved. Procedures for final disposition of unused study drug will be provided in the appropriate study manual.

#### 5.6 Prior and Concomitant Medications and/or Procedures

#### 5.6.1 Excluded Medications and/or Procedures

Participants must not receive treatment with other investigational products or devices within 30 days or 5 half-lives, whichever is longer, prior to screening.

Participants must abstain from taking any PCSK9 inhibitor within 10 weeks prior to randomization or bempedoic acid within 2 weeks prior to randomization.

#### 5.6.2 Allowed Medications and/or Procedures

Participants must be currently receiving high-intensity statin therapy (atorvastatin 40 or 80 mg or rosuvastatin 20 or 40 mg) at a stable dose for 8 weeks prior to screening and intending to remain at the same stable dose throughout the study duration.

#### 5.6.3 Documentation of Prior and Concomitant Medication Use

Medications used within 28 days prior to the Screening Visit will be recorded. Any medications administered in addition to the study drugs, whether allowed per the protocol or not, must be documented on the concomitant medication eCRF.

# 6 STUDY PROCEDURES

Study procedures will follow the Schedule of Procedures (Appendix A).

## 7 EFFICACY AND PHARMACOKINETIC ASSESSMENTS

# 7.1 Efficacy Assessments

The primary efficacy endpoint is the percent change from Day 1 to Day 84 in LDL-C for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group.

The secondary efficacy endpoints include the following, in hierarchical order:

- Percent change from Day 1 to Day 84 in LDL-C for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group;
- Percent change from Day 1 to Day 84 in ApoB for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group; and
- Percent change from Day 1 to Day 84 in ApoB for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group.

The exploratory efficacy endpoints include the following:

- Percent change from Day 1 to Day 84 in non-HDL-C, VLDL-C, HDL-C, TG, ApoE, Lp(a), and HDL-ApoE for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group and for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group; and
- Proportion of participants at Day 84 that achieve LDL-C <2.6 mmol/L (<100 mg/dL), LDL-C <1.8 mmol/L (<70 mg/dL), and LDL-C <1.3 mmol/L (<50 mg/dL) for the obicetrapib 10 mg + ezetimibe 10 mg combination treatment group compared with the placebo group and for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group.</li>

Blood samples for the lipid profile must be obtained under fasting conditions (ie, after the participant has fasted for approximately 10 hours). For the purposes of this study, fasting will be defined as nothing by mouth except water and any essential medications. If a participant is not fasting, the Investigator should reschedule the visit as soon as possible. LDL-C level will be calculated using the Friedewald equation unless  $TG \ge 400 \text{ mg/dL}$  or LDL-C  $\le 50 \text{ mg/dL}$ ; in both cases, LDL-C level will be measured directly by preparative ultracentrifugation, also referred to as beta quantification. Additionally, LDL-C will be measured by preparative ultracentrifugation, also referred to as beta quantification, at baseline (Visit 2) and at the end of the 12-week Treatment Period (Visit 4) for all participants.

#### 7.2 Pharmacokinetic Assessments

Plasma obicetrapib concentrations, both in combination with ezetimibe and as monotherapy, will be assessed at the scheduled PK collection times as indicated in Appendix A. At visits with dosing scheduled (ie, Visits 2, 3, and 4), PK samples will be collected with fasting laboratory samples (pre-dose). At Visits 3 and 4, the time between the last dose of study drug and PK sampling will be >24 hours. The subsequent post-dose PK sample at Visit 5 should be collected at approximately the same time as the previous visits.

# 7.3 Serum Archive Sample

A serum archive sample will be obtained at visits specified in the Schedule of Procedures (Appendix A) and stored for future analysis. If the sample is analyzed, it will be for non-genetic tests.

#### 8 SAFETY ASSESSMENTS

The safety and tolerability profile of obicetrapib 10 mg, both in combination with ezetimibe 10 mg and as monotherapy, will be assessed by clinical laboratory assessments (chemistry and hematology), vital signs, physical examinations, and the incidence of AEs.

#### **8.1** Adverse Events

An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and/or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational medicinal product, whether or not related to the investigational medicinal product. All AEs, including observed or volunteered problems, complaints, or symptoms, are to be recorded on the appropriate eCRF.

AEs, which include clinical laboratory assessment variables, will be monitored and documented from the time of first dose of study treatment until completion of Visit 5. Participants should be instructed to report any AE that they experience to the Investigator, whether or not they think the event is due to study drug. Beginning at the date of the first dose of study treatment, Investigators should make an assessment for AEs at each visit and record the event on the appropriate AE eCRF.

Wherever possible, a specific disease or syndrome rather than individual associated signs and symptoms should be identified by the Investigator and recorded on the eCRF. However, if an observed or reported sign or symptom is not considered a component of a specific disease or syndrome by the Investigator, it should be recorded as a separate AE on the eCRF. Additionally, the condition that led to a medical or surgical procedure (eg, surgery, endoscopy, tooth extraction, or transfusion) should be recorded as an AE, not the procedure itself.

Any medical condition already present at the date of the first dose of study treatment should be recorded as medical history and not be reported as an AE unless the medical condition or signs or symptoms present at baseline changes in severity, frequency, or seriousness at any time during the study. In this case, it should be reported as an AE.

Clinically significant abnormal laboratory or other examination findings (eg, ECG) that are detected during the study or are present at the date of the first dose of study treatment and significantly worsen during the study should be reported as AEs, as described below. The Investigator will exercise his or her medical and scientific judgment in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant. Clinically significant abnormal laboratory values occurring during the study will be followed until repeat tests return to normal, stabilize, or are no longer clinically significant. Abnormal test results that are determined to be an error should not be reported as an AE. Laboratory abnormalities or other abnormal clinical findings (eg, ECG abnormalities) should be reported as an AE if any of the following are applicable:

- If an intervention is required as a result of the abnormality;
- If action taken with the study drug is required as a result of the abnormality; or
- Based on the clinical judgment of the Investigator.

## 8.1.1 Adverse (Drug) Reaction

All noxious and unintended responses to a medicinal product related to any dose should be considered an adverse drug reaction. "Responses" to a medicinal product means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility, ie, the relationship cannot be ruled out.

# 8.1.2 Unexpected Adverse Drug Reaction

An Unexpected Adverse Drug Reaction is defined as an adverse reaction, the nature or severity of which is not consistent with the applicable product information.

## 8.1.3 Assessment of Adverse Events by the Investigator

The Investigator will assess the severity (intensity) of each AE as mild, moderate, or severe, and will also categorize each AE as to its potential relationship to study drug using the categories of yes or no.

# Assessment of severity

Mild – An event that is easily tolerated and generally not interfering with normal daily activities.

Moderate – An event that is sufficiently discomforting to interfere with normal daily activities.

Severe – An event that is incapacitating with inability to work or perform normal daily activities.

## Causality assessment

The relationship of an AE to the administration of the study drug is to be assessed according to the following definitions:

No (unrelated, not related, unlikely to be related) – The time course between the administration of study drug and the occurrence or worsening of the AE rules out a causal relationship and another cause (concomitant drugs, therapies, complications, etc) is suspected.

Yes (possibly, probably, or definitely related) – The time course between the administration of study drug and the occurrence or worsening of the AE is consistent with a causal relationship and no other cause (concomitant drugs, therapies, complications, etc) can be identified.

The definition implies a <u>reasonable</u> possibility of a causal relationship between the event and the study drug. This means that there are facts (evidence) or arguments to suggest a causal relationship.

The following factors should also be considered:

• The temporal sequence from study drug administration-

The event should occur after the study drug is given. The length of time from study drug exposure to event should be evaluated in the clinical context of the event.

• Underlying, concomitant, intercurrent diseases-

Each report should be evaluated in the context of the natural history and course of the disease being treated and any other disease the participant may have.

# • Concomitant drug-

The other drugs the participant is taking or the treatment the participant receives should be examined to determine whether any of them might be recognized to cause the event in question.

• Known response pattern for this class of study drug-

Clinical and/or preclinical data may indicate whether a particular response is likely to be a class effect.

Exposure to physical and/or mental stresses-

The exposure to stress might induce adverse changes in the recipient and provide a logical and better explanation for the event.

• The pharmacology and PK of the study drug-

The known pharmacologic properties (absorption, distribution, metabolism, and excretion) of the study drug should be considered.

## 8.2 Serious Adverse Events

An AE or adverse reaction is considered serious if, in the view of either the Investigator or Sponsor, it results in any of the following outcomes:

- Death:
- A life-threatening AE;

Note: An AE or adverse reaction is considered "life-threatening" if, in view of either the Investigator or Sponsor, its occurrence places the participant at <u>immediate risk</u> of death. It does not include an event that, had it occurred in a more severe form, might have caused death.

• Requires hospitalization or prolongation of existing hospitalizations;

Note: Any hospital admission with at least 1 overnight stay will be considered an inpatient hospitalization. An emergency room or urgent care visit without hospital admission will not be recorded as a SAE under this criterion, nor will hospitalization for a procedure scheduled or planned before signing of informed consent, or elective treatment of a pre-existing condition that did not worsen from baseline. However, unexpected complications and/or prolongation of hospitalization that occur during elective surgery should be recorded as AEs and assessed for seriousness. Admission to the hospital for social or situational reasons (ie, no place to stay, live too far away to come for hospital visits, respite care) will not be considered inpatient hospitalizations.

- A persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions;
- A congenital anomaly/birth defect; or
- An important medical event.

Note: Important medical events that do not meet any of the above criteria may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent 1 of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment
in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalizations, or the development of drug dependency.

# 8.3 Serious Adverse Event Reporting – Procedures for Investigators

# **Initial reports**

All SAEs occurring from the time of the first dose of study treatment until 30 days following the last administration of study drug must be reported to within 24 hours of the knowledge of the occurrence. After the 30-day reporting window, any SAE that the Investigator considers related to study drug must be reported to sponsor/designee.

To report the SAE, complete the SAE form electronically in the electronic data capture (EDC)

system for the study. When the form is completed, personnel will be notified electronically by the EDC system and will retrieve the form. If the event meets serious criteria and it is not possible to access the EDC system, send an email to at or call the reporting line (phone number listed below), and fax/email the completed paper SAE form to (contact information listed in Section 8.6) within 24 hours of awareness. When the EDC system becomes available, the SAE information must be entered within 24 hours of the system becoming available.

## Follow-up reports

The Investigator must continue to follow the participant until the SAE has subsided or until the condition becomes chronic in nature, stabilizes (in the case of persistent impairment), or the participant dies.

Within 24 hours of receipt of follow-up information, the Investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, participant discharge summary or autopsy reports) to via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

## 8.4 Pregnancy Reporting

If a participant becomes pregnant during the study or within the Safety Follow-up Period defined in the protocol, the Investigator is to stop dosing with study drug(s) immediately and the participant should be withdrawn from the study. Early termination procedures should be implemented at that time.

| A pregna | ancy | is not considered | to b | e an AE or | SA | E; how | ever, it | must b | e rep | ported to | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | within 24 hour | s of | knowledge | of t | he ever | nt. | | | wil | 1 then |
| provide | the | Investigator/site | the | Exposure | In | Utero | (EIU) | form | for | completion. | The |
| Investiga | ator/s | ite must complete | the l | EIU form aı | nd fa | x/email | l it back | to | | | |

If the female partner of a male participant becomes pregnant while the participant is receiving study drug or within the Safety Follow-up Period defined in the protocol, the Investigator should notify as described above.

The pregnancy should be followed until the outcome of the pregnancy, whenever possible. Once the outcome of the pregnancy is known, the EIU form should be completed and faxed/emailed to

. If the outcome of the pregnancy meets the criteria for immediate classification as an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), the Investigator should follow the procedures for reporting an SAE.

## 8.5 Expedited Reporting

The Sponsor/designee will report all relevant information about Suspected Unexpected Serious Adverse Reactions (SUSARs) that are fatal or life-threatening as soon as possible to the FDA, and in any case no later than 7 days after knowledge by the Sponsor/designee of such a case. Relevant follow-up information will subsequently be communicated within an additional 8 days.

All other SUSARs will be reported to the FDA, applicable competent authorities concerned, and to the Central Ethics Committee concerned as soon as possible but within a maximum of 15 days of first knowledge by the Sponsor/designee.

The Sponsor/designee will also report any additional expedited safety reports required in accordance with the timelines outlined in country-specific legislation.

The Sponsor/designee will also inform all Investigators as required per local regulation.

The requirements above refer to the requirements relating to study drug.

## **8.6** Special Situation Reports

Special situation reports include reports of overdose, misuse, abuse, medication error, and reports of adverse reactions associated with product complaints.

- Overdose: Refers to the administration of a quantity of a medicinal product given per administration or cumulatively (accidentally or intentionally), which is above the maximum recommended dose according to the protocol. Clinical judgement should always be applied. In cases of a discrepancy in the drug accountability, overdose will be established only when it is clear that the participant has taken additional dose(s) or the Investigator has reason to suspect that the participant has taken additional dose(s).
- **Misuse:** Refers to situations where the medicinal product is intentionally and inappropriately used not in a way that is not in accordance with the protocol instructions or local prescribing information and may be accompanied by harmful physical and/or psychological effects.
- **Abuse:** Is defined as persistent or sporadic, intentional excessive use of a medicinal product, which is accompanied by harmful physical or psychological effects.
- **Medication error:** Is any unintentional error in the prescribing, dispensing, or administration of a medicinal product by a healthcare professional, participant, or consumer, respectively. The administration or consumption of the unassigned treatment and administration of an expired product are always reportable as medication errors, cases of participants missing doses of investigational product are not considered reportable as medication error.
- **Product complaint:** Is defined as any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, or performance of a drug or device after it is released for distribution. A special situations form will only be completed if a complaint is associated with an adverse drug reaction.

All special situation events as described above must be reported on the Special Situations Report form and faxed/emailed to (contact information listed below) within 24 hours of knowledge of the event. All AEs associated with these Special Situation reports should be reported as AEs or SAEs as well as recorded on the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome should be provided, when available.



## 8.7 Clinical Laboratory Evaluations

## 8.7.1 Chemistry and Hematology Assessments

Blood for chemistry and hematology will be obtained as indicated in Appendix A and sent to a central laboratory for analysis. See Appendix B for a complete list of analytes. Blood samples for chemistry and hematology must be obtained under fasting conditions (ie, after the participant has fasted for approximately 10 hours). For the purposes of this study, fasting will be defined as nothing by mouth except water and any essential medications. If a participant is not fasting, the Investigator should reschedule the visit as soon as possible. Estimated glomerular filtration rate will be calculated using the Chronic Kidney Disease Epidemiology Collaboration equation. At the Screening Visit only, the chemistry panel will include HbA1c.

## 8.7.2 Endocrinology Assessments

A urine pregnancy test will be performed for women of childbearing potential at the Screening Visit prior to their participation in the study and at the Early Termination Visit (if indicated).

An FSH test will be performed at the Screening Visit prior to participation in the study in women <55 years of age for whom it has been ≥1 year since their last menstrual period.

#### 8.7.3 Aldosterone Assessment

A plasma sample for aldosterone will be collected at visits specified in the Schedule of Procedures (Appendix A). Samples must be obtained under fasting conditions (ie, after the participant has fasted for approximately 10 hours).

#### 8.8 Vital Signs

Vital signs will be taken as indicated in Appendix A. Vital signs will include body temperature, heart rate, and triplicate blood pressure (systolic and diastolic) measurements. Participants should be in the supine position after at least 10 minutes rest prior to the vital sign measurements.

# 8.9 Weight and Height

Weight and height will be measured at the Screening Visit and will be used to calculate body mass index. Measurement of weight should be performed with the participant dressed in indoor clothing, with shoes removed, and bladder empty.

# 8.10 Demographics

Participant demographic data (eg, gender, race, ethnicity, and birth date/year) will be collected at the Screening Visit.

# 8.11 Electrocardiograms

A single, standard 12-lead ECG will be performed by the Investigator or trained site personnel at the Screening Visit and read locally.

# 8.12 Physical Examinations

A physical examination will be performed as indicated in Appendix A.

## 9 STATISTICS

## 9.1 Analysis Populations

The Intent-to-Treat (ITT) Population will include all participants randomized into the study. Treatment classification will be based on the randomized treatment.

The Modified ITT (mITT) Population will include all participants in the ITT Population who receive at least 1 dose of any study drug and have a baseline value for the LDL-C assessment. Any efficacy measurement obtained during the Safety Follow-up Visit (Visit 5) after a participant permanently discontinues the study drug or after a participant receives an excluded medication and/or procedure will be removed from the mITT analysis. Treatment classification will be based on the randomized treatment. The mITT Population will be used for the primary analysis of all efficacy endpoints.

The Per-Protocol (PP) Population will include all participants in the mITT Population who have a baseline value for the LDL-C assessment, have a Day 84 value for the LDL-C assessment, and who do not experience a major protocol deviation that could potentially impact the primary efficacy endpoint. The PP Population, along with the reason for exclusion, will be finalized prior to study unblinding.

The PK Population will include all participants in the mITT Population who have sufficient blood samples collected for valid estimation of PK parameters.

The Safety Population will include all participants who receive at least 1 dose of any study drug. Treatment classification will be based on the actual treatment received. The Safety Population will be the primary population used for the safety analyses.

## 9.2 Statistical Methods

A Statistical Analysis Plan (SAP) will be finalized before database lock. Any changes to the methods described in the SAP will be described and justified as needed in the Clinical Study Report. All study-collected data will be summarized by treatment group using descriptive statistics, graphs, and/or raw data listings. Descriptive statistics for continuous variables will include number of participants (n), mean, standard deviation (SD), median, minimum, and maximum values. Analysis of categorical variables will include frequency and percentage.

## 9.2.1 Analysis of Efficacy

The mITT Population will be the primary population for the efficacy analyses. Efficacy will also be analyzed using the ITT Population and the PP Population as supportive analyses.

## 9.2.1.1 Primary efficacy analysis

The primary efficacy analysis of the percent change from Day 1 to Day 84 in LDL-C will be performed using a mixed model for repeated measures (MMRM) approach. The analysis will include fixed effects for treatment, visit, and treatment-by-visit interaction, along with a covariate of the baseline value as a continuous covariate. The Restricted Maximum Likelihood estimation approach will be used with an unstructured covariance matrix. The least squares means, standard errors, and 2-sided 95% confidence intervals for the combination group and for comparison of the combination treatment group to the placebo group will be provided. Sensitivity analyses for various assumptions of missing data will be imputed using multiple imputation methodology.

Results will be combined using Rubin's method. Full details of the model(s) and imputation will be provided in the SAP.

## 9.2.1.2 Secondary efficacy analyses

Similar MMRM models will be developed to examine the secondary efficacy endpoints. In order to maintain the overall Type I error rate, the secondary efficacy endpoints will be tested sequentially at the 0.05 significance level according to the order of hierarchy specified in Section 7.1.

## 9.2.1.3 Exploratory analyses

Similar MMRM models will be used for the percent change from Day 1 to Day 84 in non-HDL-C, VLDL-C, HDL-C, TG, ApoE, Lp(a), and HDL-ApoE.

The proportion of participants at Day 84 that achieve LDL-C <2.6 mmol/L (<100 mg/dL), LDL-C <1.8 mmol/L (<70 mg/dL), and LDL-C <1.3 mmol/L (<50 mg/dL) will be examined through logistic regression models for binary variables with covariants of the treatment groups and the baseline variable.

No adjustment will be made for multiplicity in testing the exploratory efficacy endpoints. Nominal p-values will be provided when applicable. Any additional sensitivity and/or supplemental analyses will be defined in the SAP.

## 9.2.2 Analysis of Pharmacokinetics

Plasma obicetrapib concentrations will be summarized with descriptive statistics based on the PK Population. Exploration of any relationships with obicetrapib exposure will be performed, as appropriate.

# 9.2.3 Analysis of Safety

The Safety Population will be the primary population for the safety analyses. All safety endpoints will be summarized descriptively. No statistical inference will be applied to the safety endpoints.

AEs will be categorized by primary system organ class and preferred term as coded using the Medical Dictionary for Regulatory Activities category designations. Summaries of AEs, including the number and percentage of participants who experience an AE, will be provided.

Laboratory values will be summarized descriptively, including the change from baseline, by treatment group, and overall. In addition, shift tables will be presented to describe the change in laboratory parameter values at post-baseline visits using normal range categories (low, normal, and high).

## 9.2.4 Interim Analysis

No interim analysis is planned for this study.

## 9.2.5 Sample Size Determination

A sample size of at least 108 evaluable participants (ie, 36 participants per treatment group) will provide >90% power to detect a 30% difference in LDL-C reduction at Day 84 (SD of 15%) for each of the obicetrapib treatment groups compared with the placebo group at a 1-sided significance level of 0.025.

The sample size for this study was determined in order to provide sufficient power for the analyses of the primary and first secondary efficacy endpoints described in Section 7.1. Therefore, assuming an approximately 5% dropout rate, enrollment of approximately 114 participants (ie, 38 participants per treatment group) is planned for this study. This sample size will also contribute sufficient participant exposure and safety data.

Participants will be stratified according to their Screening Visit LDL-C levels ( $\geq 100 \text{ or } < 100 \text{ mg/dL}$ ).

#### 10 DATA MANAGEMENT AND RECORD KEEPING

## 10.1 Data Management

## 10.1.1 Data Handling

Data will be recorded at the site on eCRFs and reviewed by the Clinical Research Associate (CRA) during monitoring visits. The CRAs will verify data recorded in the EDC system with source documents. All corrections or changes made to any study data must be appropriately tracked in an audit trail in the EDC system. An eCRF will be considered complete when all missing, incorrect, and/or inconsistent data has been accounted for.

# 10.1.2 Computer Systems

Data will be processed using a validated computer system conforming to regulatory requirements.

## 10.1.3 Data Entry

Data must be recorded using the EDC system as the study is in progress. All site personnel must log into the system using their secure username and password in order to enter, review, or correct study data. These procedures must comply with Title 21 of the Code of Federal Regulations Part 11 and other appropriate international regulations. All passwords will be strictly confidential.

# 10.1.4 Medical Information Coding

For medical information, the following thesauri will be used:

- Medical Dictionary for Regulatory Activities (latest) for medical history and AEs; and
- WHO Drug Dictionary for prior and concomitant medications.

## 10.1.5 Data Validation

Validation checks programmed within the EDC system, as well as supplemental validation performed via review of the downloaded data, will be applied to the data in order to ensure accurate, consistent, and reliable data. Data identified as erroneous, or data that are missing, will be referred to the site for resolution through data queries.

The eCRFs must be reviewed and electronically signed by the Investigator.

# 10.2 Record Keeping

Records of participants, source documents, monitoring visit logs, eCRFs, inventory of study drug, regulatory documents, and other Sponsor correspondence pertaining to the study must be kept in the appropriate study files at the site. Source data are defined as all information in original records and certified copies of original records of clinical findings, observations, or other activities in a clinical study necessary for the evaluation and reconstruction of the clinical study. Source data are contained in source documents (original records or certified copies). These records will be retained in a secure file for the period as set forth in the Clinical Study Agreement. Prior to transfer or destruction of these records, the Sponsor must be notified in writing and be given the opportunity to further store such records.

# 10.3 End of Study

The end of the study ("study completion") is defined as the date of the last protocol-specified visit/assessment (including telephone contact) for the last participant in the study.

# 11 INVESTIGATOR REQUIREMENTS AND QUALITY CONTROL

## 11.1 Ethical Conduct of the Study

Good Clinical Practice (GCP) is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve human participants. Compliance with this standard provides public assurance that the rights, safety, and wellbeing of study participants are protected, consistent with the principles that have their origin in the Declaration of Helsinki, and that the clinical study data are credible.

#### 11.2 Institutional Review Board

The Institutional Review Board (IRB) will review all appropriate study documentation in order to safeguard the rights, safety, and well-being of participants. The study will only be conducted at sites where IRB approval has been obtained. The protocol, Investigator's Brochure, ICF, advertisements (if applicable), written information given to the participants, safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB by the Investigator.

Federal regulations and ICH Guidelines require that approval be obtained from an IRB prior to participation of participants in research studies. Prior to study onset, the protocol, any protocol amendments, ICFs, advertisements to be used for participant recruitment, and any other written information regarding this study to be provided to a participant or participant's legal guardian must be approved by the IRB.

No study drug will be released to the site for dosing until written IRB authorization has been received by the Sponsor.

## 11.3 Informed Consent

The ICF and any changes to the ICF made during the course of the study must be agreed to by the Sponsor or designee and the IRB prior to its use and must be in compliance with all ICH GCP, local regulatory requirements, and legal requirements.

The Investigator must ensure that each study participant is fully informed about the nature and objectives of the study and possible risks associated with participation and must ensure that the participant has been informed of his/her rights to privacy. The Investigator will obtain written informed consent from each participant before any study-related activity is performed and should document in the source documentation that consent was obtained prior to enrollment in the study. The original signed copy of the ICF must be maintained by the Investigator and is subject to inspection by a representative of the Sponsor, their representatives, auditors, the IRB, and/or regulatory agencies. A copy of the signed ICF will be given to the participant.

## 11.4 Study Monitoring Requirements

It is the responsibility of the Investigator to ensure that the study is conducted in accordance with the protocol, Declaration of Helsinki, ICH GCP, and applicable regulatory requirements, and that valid data are entered into the eCRFs.

To achieve this objective, the CRA's duties are to aid the Investigator and, at the same time, the Sponsor in the maintenance of complete, legible, well organized, and easily retrievable data. Before the enrollment of any participant in this study, the Sponsor or their designee will review

with the Investigator and site personnel the following documents: protocol, Investigator's Brochure, eCRFs and procedures for their completion, informed consent process, and the procedure for reporting SAEs.

The Investigator will permit the Sponsor or their designee to monitor the study as frequently as deemed necessary to determine that data recording and protocol adherence are satisfactory. During the monitoring visits, information recorded on the eCRFs will be verified against source documents and requests for clarification or correction may be made. After the eCRF data is entered by the site, the CRA will review the data for safety information, completeness, accuracy, and logical consistency. Computer programs that identify data inconsistencies may be used to help monitor the clinical study. If necessary, requests for clarification or correction will be sent to Investigators. The Investigator and his/her staff will be expected to cooperate with the Sponsor or their designee and provide any missing information, whenever possible.

All monitoring activities will be reported and archived. In addition, monitoring visits will be documented at the investigational site by signature and date on the study-related monitoring log.

#### 11.5 Disclosure of Data

Data generated by this study must be available for inspection by the FDA, the Sponsor or their designee, applicable foreign health authorities, and the IRB as appropriate. Participants or their legal representatives may request their medical information be given to their personal physician or other appropriate medical personnel responsible for their welfare.

Participant medical information obtained during the study is confidential and disclosure to third parties other than those noted above is prohibited.

#### 11.6 Retention of Records

To enable evaluations and/or audits from regulatory authorities or the Sponsor, the Investigator will keep records, including the identity of all participants (sufficient information to link records, eg, eCRFs and hospital records), all original signed ICFs, copies of all eCRFs, SAE forms, source documents, and detailed records of treatment disposition. The records should be retained by the Investigator according to specifications in the ICH guidelines, local regulations, or as specified in the Clinical Study Agreement, whichever is longer. The Investigator must obtain written permission from the Sponsor before disposing of any records, even if retention requirements have been met.

If the Investigator relocates, retires, or for any reason withdraws from the study, the Sponsor should be prospectively notified. The study records must be transferred to an acceptable designee, such as another Investigator, another institution, or to the Sponsor.

## 11.7 Publication Policy

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. Each Investigator is obligated to keep data pertaining to the study confidential. The Investigator must consult with the Sponsor before any study data are submitted for publication. The Sponsor reserves the right to deny publication rights until mutual agreement on the content, format, interpretation of data in the manuscript, and journal selected for publication are achieved.

## 11.8 Financial Disclosure

Investigators are required to provide financial disclosure information to the Sponsor to permit the Sponsor to fulfill its obligations under 21 Code of Federal Regulations Part 54. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of 1 year after the completion of the study.

## 12 STUDY ADMINISTRATIVE INFORMATION

## 12.1 Protocol Amendments

Any amendments to the study protocol will be communicated to the Investigators by the Sponsor. All protocol amendments will undergo the same review and approval process as the original protocol. A protocol amendment may be implemented after it has been approved by the IRB, unless immediate implementation of the change is necessary for participant safety. In this case, the situation must be documented and reported to the IRB within 5 working days.

#### 13 REFERENCES

- 1. de Grooth GJ, Klerkx AH, Stroes ES, et al. A review of CETP and its relation to atherosclerosis. *J Lipid Res.* 2004;45(11):1967-1974.
- 2. Ference BA, Kastelein JJ, Ginsberg HN, et al. Association of genetic variants related to CETP inhibitors and statins with lipoprotein levels and cardiovascular risk. *JAMA*. 2017;318(10):947-956.
- 3. Tall AR, Rader DJ. Trials and tribulations of CETP inhibitors. *Circ Res.* 2018;122(1):106-112.
- 4. Ference BA, Kastelein JJP, Ray KK, et al. Association of triglyceride-lowering LPL variants and LDL-C-lowering LDLR variants with risk of coronary heart disease. *JAMA*. 2019;321(4):364-373.
- 5. Hovingh GK, Kastelein JJ, van Deventer SJ, et al. Cholesterol ester transfer protein inhibition by TA-8995 in patients with mild dyslipidaemia (TULIP): a randomised, double-blind, placebo-controlled phase 2 trial. *Lancet*. 2015;386(9992):452-460.
- 6. van Capelleveen JC, Kastelein JJ, Zwinderman AH, et al. Effects of the cholesteryl ester transfer protein inhibitor, TA-8995, on cholesterol efflux capacity and high-density lipoprotein particle subclasses. *J Clin Lipidol*. 2016;10(5):1137-1144.e3.
- 7. Cholesterol Treatment Trialists' (CTT) Collaboration. Baigent C, Blackwell L, Emberson J, et al. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. *Lancet*. 2010;376(9753):1670-1681.
- 8. Pandor A, Ara RM, Tumur I, et al. Ezetimibe monotherapy for cholesterol lowering in 2,722 people: systematic review and meta-analysis of randomized controlled trials. *J Intern Med.* 2009;265(5):568-580.
- 9. Morrone D, Weintraub WS, Toth PP, et al. Lipid-altering efficacy of ezetimibe plus statin and statin monotherapy and identification of factors associated with treatment response: a pooled analysis of over 21,000 subjects from 27 clinical trials. *Atherosclerosis*. 2012;223(2):251-261.
- 10. Cannon CP, Blazing MA, Giugliano RP, et al. Ezetimibe added to statin therapy after acute coronary syndromes. *N Engl J Med*. 2015;372(25):2387-2397.
- 11. United States Food and Drug Administration. FDA guidance on conduct of clinical trials of medical products during the COVID-19 public health emergency. *Guidance for Industry, Investigators, and Institutional Review Boards.* March 2020, updated 27 January 2021. https://www.fda.gov/media/136238/download. Accessed 04 August 2021.
- 12. Levey AS. CKD-EPI equations for glomerular filtration rate (GFR). MDCalc. https://www.mdcalc.com/ckd-epi-equations-glomerular-filtration-rate-gfr. Accessed 09 November 2020.
- 13. Friedewald W. LDL calculated. MDCalc. https://www.mdcalc.com/ldl-calculated. Accessed 10 August 2021.

# **APPENDIX A: SCHEDULE OF PROCEDURES**

| | Screening <sup>a,b</sup> | Treatment Period | | | Safety Follow-Up | |
|---|---|---|---|---|---|---|
| Visit | 1 | 2 (Baseline) | 3 | 4 (EOT) | 5 | |
| Week | Up to -2 | 0 | 4 | 12 | 16 | Early Termination Visit |
| Day (±Visit Window) | -14 to -1 | 1 | 28 (±2) | 84 (±2) | 112 (±2) | Unscheduled |
| Informed consent <sup>c</sup> | X | | | | | |
| Inclusion/exclusion criteria | X | $X^d$ | | | | |
| Demographic information | X | | | | | |
| Medical/surgical history | X | | | | | |
| Prior/concomitant medications | X | X | X | X | X | X |
| Weight and height <sup>e</sup> | X | | | | | |
| Physical examination | X | | | X | | |
| Vital signs <sup>f</sup> | X | X | X | X | X | X |
| 12-lead ECG <sup>g</sup> | X | | | | | |
| Urine pregnancy test <sup>h</sup> | X | | | | | X |
| FSH test <sup>i</sup> | X | | | | | |
| Fasting (approximately 10 hours) | | | | | | |
| chemistry and hematology <sup>j</sup> | X | X | X | X | X | X |
| Fasting (approximately 10 hours) | | | | | | |
| lipid profile <sup>k</sup> | X | X | X | X | | X |
| PK sample <sup>1</sup> | | X | X | X | X <sup>m</sup> | X |
| Fasting (approximately 10 hours) | | | | | | |
| aldosterone | | X | X | X | X | X |
| Fasting (approximately 10 hours) | | | | | | |
| Lp(a) | | X | | X | | |
| Serum archive sample <sup>n</sup> | | X | | X | | |
| Randomization | | X | | | | |
| Dispense study drug <sup>o</sup> | | X | X | | | |
| Study drug administration <sup>p</sup> | | | X | | | |
| Study drug compliance | | | X | X | | |
| Register visit in IRT | X | X | X | X | | X |
| Adverse events | | X | X | X | X | X |

Note: When several assessments are required at the same visit, samples for clinical laboratory assessments should be collected after completing other assessments, such as physical examinations, vital signs, and 12-lead ECGs.

Note: In cases of COVID-19 limitations, it is the Investigator's responsibility to assure the safety of participants. If necessary, the Sponsor will implement and document mitigation strategies as described in Section 3.1.4. In the absence of a COVID-19 impact, it is expected that Investigators and participants follow the protocol requirements as set forth.

Note: For the purposes of this study, fasting will be defined as nothing by mouth except water and any essential medications.

- a. If laboratory abnormalities during screening are considered by the Investigator to be transient, then the laboratory tests may be repeated once during screening. The Investigator's rationale for retesting should be documented. If the retest result is no longer exclusionary, the participant may be randomized.
- b. A participant who is screened and does not meet the study eligibility criteria may be considered for rescreening upon Sponsor and/or Medical Monitor consultation and approval. Rescreened participants will be assigned a new participant number. Rescreening should occur no less than 5 days after the last Screening Visit.
- c. Participants will be required to sign an ICF before any study-related procedures are performed.
- d. Confirm the participant continues to meet the inclusion and exclusion criteria and assess any updates since the Screening Visit.
- e. Weight and height will be measured at the Screening Visit and will be used to calculate body mass index. Measurement of weight should be performed with the participant dressed in indoor clothing, with shoes removed, and bladder empty.
- f. Vital signs will include body temperature, heart rate, and triplicate blood pressure (systolic and diastolic) measurements. Participants should be in the supine position after at least 10 minutes rest prior to the vital sign measurements.
- g. A single, standard 12-lead ECG will be performed by the Investigator or trained site personnel at the Screening Visit and read locally.
- h. For women of childbearing potential only.
- i. FSH test will be performed in women <55 years of age for whom it has been ≥1 year since their last menstrual period.
- j. At the Screening Visit only, chemistry panel will include HbA1c.
- k. LDL-C level will be calculated using the Friedewald equation unless TG≥400 mg/dL or LDL-C ≤50 mg/dL; in both cases, LDL-C level will be measured directly by preparative ultracentrifugation, also referred to as beta quantification (Source: LDL calculated. MDCalc. https://www.mdcalc.com/ldl-calculated. Accessed 10 August 2021). Additionally, LDL-C will be measured by preparative ultracentrifugation, also referred to as beta quantification, at baseline (Visit 2) and at the end of the 12-week Treatment Period (Visit 4) for all participants.
- 1. At visits with dosing scheduled (ie, Visits 2, 3, and 4), PK samples will be collected with fasting laboratory samples (pre-dose). At Visits 3 and 4, the time between the last dose of study drug and PK sampling will be >24 hours. The subsequent post-dose PK sample at Visit 5 should be collected at approximately the same time as the previous visits.
- m. PK samples will not be collected during the Safety Follow-up Visit for participants who discontinue study drug early without withdrawing consent or for participants who withdraw prematurely from the study.
- n. A serum archive sample will be obtained and stored for future analysis. If the sample is analyzed, it will be for non-genetic tests.
- o. At Visit 2 (Day 1), participants will receive 1 kit (containing 32 obicetrapib tablets or matching placebo tablets and 32 ezetimibe capsules or matching placebo capsules totaling 64 tablets/capsules per kit) with the study drugs appropriate for the participant's treatment group. At Visit 3 (Day 28), participants will receive 2 kits as described above. Each kit will provide a sufficient supply for 28 days of dosing, with enough for an extra 4 days of dosing in case the participant needs to postpone the next visit. Participants will be instructed to take 2 units from the kit each day. The kit will be clearly labelled to indicate which tablets/capsules to use on each day. Participants will be instructed to bring all unused study drugs to the site at the next visit.
- p. Study drugs (1 tablet and 1 capsule) will be administered by the participant orally with water, once daily on Day 1 to Day 84 at approximately the same time each morning. On days with visits scheduled, study drugs should be administered with water following all fasted blood samples. At Visits 3 and 4, participants will dose from the kit received at the previous visit (Visits 2 and 3, respectively).

COVID-19 = Coronavirus Disease 2019; ECG = electrocardiogram; EOT = End of Treatment; FSH = follicle-stimulating hormone; HbA1c = glycosylated hemoglobin; ICF = informed consent form; IRT = interactive response technology; LDL-C = low-density lipoprotein cholesterol; Lp(a) = lipoprotein (a); PK = pharmacokinetic; TG = triglyceride(s).

## APPENDIX B: CLINICAL LABORATORY ANALYTES

# **Standard Safety Chemistry Panel**

Alanine aminotransferase Albumin
Alkaline phosphatase Amylase
Aspartate aminotransferase Bicarbonate
Blood urea nitrogen Calcium

Chloride Creatine kinase

Creatinine Estimated glomerular filtration rate [1]

Gamma-glutamyl transferase Glucose (fasting)

Glycosylated hemoglobin [2] High-sensitivity C-reactive protein

Inorganic phosphorus Lactate dehydrogenase

Lipase Potassium
Sodium Total bilirubin
Total protein Uric acid

 Calculated using the Chronic Kidney Disease Epidemiology Collaboration equation. (Source: CKD-EPI equations for glomerular filtration rate [GFR]. MDCalc. https://www.mdcalc.com/ckd-epi-equations-glomerular-filtration-rate-gfr. Accessed 09 November 2020).

Screening Visit only.

## **Endocrinology**

Aldosterone Follicle-stimulating hormone [1]

Urine pregnancy test [2]

- 1. Follicle-stimulating hormone test will be performed in women <55 years of age for whom it has been ≥1 year since their last menstrual period.
- 2. For women of childbearing potential only.

## Hematology

Hematocrit Hemoglobin

Platelets Red blood cell count

White blood cell count and differential [1]

 Manual microscopic review is performed only if white blood cell count and/or differential values are out of reference range.

## **Lipid Profile**

Apolipoprotein B Apolipoprotein E (Apo E)

High-density lipoprotein-ApoE High-density lipoprotein cholesterol
Low-density lipoprotein cholesterol [1] Non-high-density lipoprotein cholesterol
Triglycerides Very low-density lipoprotein cholesterol

1. LDL-C will be calculated using the Friedewald equation unless triglycerides ≥400 mg/dL or low-density lipoprotein cholesterol (LDL-C) ≤50 mg/dL; in both cases, LDL-C level will be measured directly by preparative ultracentrifugation, also referred to as beta quantification (Source: LDL calculated. MDCalc. https://www.mdcalc.com/ldl-calculated. Accessed 10 August 2021). In addition, for all participants, LDL-C will be measured by preparative ultracentrifugation, also referred to as beta quantification, at baseline (Visit 2) and at the end of the 12-week Treatment Period (Visit 4).

# **Other Laboratory Analytes**

Lipoprotein (a)